CLINICAL TRIAL: NCT04257617
Title: First in Human, Phase I Trial of ZL-1201 in Subjects With Advanced Cancer
Brief Title: A Trial of ZL-1201 in Subjects With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zai Lab (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Zai Lab (Hong Kong), Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZL-1201-001
Record Dates: First submitted 2020-01-27; First posted 2020-02-06 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-02

CONDITIONS: Advanced Cancer
Keywords: Advanced solid tumors or hematologic malignancies
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Single arm, ZL-1201 (Experimental): Single arm, ZL-1201
  Interventions: Drug: ZL-1201

INTERVENTIONS:
Drug: ZL-1201 — Part 1 & 2: Escalating dose of ZL-1201, Part 3: three dose levels determined from Part 1 and Part 2.
  Other Names: Monotherapy

SUMMARY:
First in Human, Phase I Trial of ZL-1201 in Subjects with Advanced Cancer

DETAILED DESCRIPTION:
This is a first-in-human, dose escalation trial of ZL-1201. The major aims of the study are to define the safety profile of this new drug, and to determine a recommended dose and schedule for potential additional trials.

ELIGIBILITY:
Inclusion Criteria:

* Histologically/cytologically confirmed, locally advanced unresectable or metastatic solid tumors and lymphomas that are refractory or intolerant to standard of care therapy, or for which no standard therapy exists.
* Adequate hematologic status
* Adequate coagulation function
* Adequate hepatic function
* Adequate renal function

Exclusion Criteria:

* Known active brain metastases
* Red blood cells transfusion dependence
* Known cardiopulmonary disease
* Pregnant or breast-feeding females
* Any other serious underlying medical

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2022-05-17 (Actual); Study Completion 2023-01-19 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of ZL-1201 when administered as an intravenous (IV) infusion: Incidence of Treatment-Emergent Adverse Events | From the time of informed consent to 30 days after last dose
  Incidence of Treatment-Emergent Adverse Events as Assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetics：AUC | Up to 30 days after last dose
  The area under the curve (AUC) of serum concentration of the drug after the administration
Pharmacokinetics: Cmax | Up to 30 days after last dose
  Maximum serum concentration(Cmax) of the drug after the administration
Pharmacokinetics: t1/2 | Up to 30 days after last dose
  Half-life(t1/2) of the drug
Pharmacokinetics: CL | Up to 30 days after last dose
  Total body clearance of the drug
Pharmacokinetics: Vss | Up to 30 days after last dose
  Volume of the distrubution at steady-state
Immunogenicity | Up to 30 days after last dose
  Anti-Drug Antibodies (ADA) will be tested and percentage of ADA positive patients will be calculated to evaluate immunogenicity
Overall Response Rate (ORR） | Up to 2 years after enrollment
  ORR includes CR and PR

CONTACTS AND LOCATIONS:
Overall Officials: Study Physician, Study Director — Zai Laboratory
Locations (7):
- United States (5):
  - US2004, Phoenix, Arizona
  - US2005, Jacksonville, Florida
  - US2001, Rochester, Minnesota
  - US2003, St Louis, Missouri
  - US2002, New York, New York
- China (2):
  - CN1003, Chongqing, Chongqing Municipality
  - CN1002, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No